CLINICAL TRIAL: NCT04704830
Title: A Phase III Randomized Controlled Multi-centre Trial to Evaluate the Efficacy of the R21/Matrix-M Vaccine in African Children Against Clinical Malaria
Brief Title: R21/Matrix-M in African Children Against Clinical Malaria
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Institut de Recherche en Sciences de la Sante, Burkina Faso (Other Government); Institut de Recherche en Sciences de la Sante-Direction Regionale de l'Ouest (Other Government); Malaria Research and Training Center, Bamako, Mali (Other); KEMRI-Wellcome Trust Collaborative Research Program (Other); Ifakara Health Institute Clinical Trial Facility, Bagamoyo Research and Training Centre, PO Box 74, Bagamoyo, Tanzania (Unknown); London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VAC078
Record Dates: First submitted 2021-01-07; First posted 2021-01-12 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — Rabies Vaccines; Hepatitis A Vaccines; Meningococcal Vaccines

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (11):
- Standard Regime - Group 1-1 (Experimental): R21/Matrix-M at primary series and first booster, control vaccine at second and third booster, n = 400, 5-36 months olds
  Interventions: Biological: R21/Matrix-M; Biological: Rabies vaccine, Hepatitis A vaccine or Meningococcal vaccine
- Standard Regime - Group 1-2 (Experimental): R21/Matrix-M at primary series, first booster and second booster, control vaccine at third booster, n = 400, 5-36 months olds
  Interventions: Biological: R21/Matrix-M; Biological: Rabies vaccine, Hepatitis A vaccine or Meningococcal vaccine
- Standard Regime - Group 1-3 (Experimental): R21/Matrix-M at primary series and first booster, control vaccine at second booster and R21/Matrix-M at third booster, n = 400, 5-36 months olds
  Interventions: Biological: R21/Matrix-M; Biological: Rabies vaccine, Hepatitis A vaccine or Meningococcal vaccine
- Standard Regime - Group 1-4 (Experimental): R21/Matrix-M at primary series, first booster, second booster and third booster, n = 400, 5-36 months olds
  Interventions: Biological: R21/Matrix-M
- Standard Regime - Group 2 (Placebo Comparator): Control vaccine at primary series, first booster, second booster and third booster, n=800, 5-36 month olds
  Interventions: Biological: Rabies vaccine, Hepatitis A vaccine or Meningococcal vaccine
- Seasonal Regime - Group 5 (Experimental): Group 3-1 for the initial part of the trial and first extension - R21/Matrix-M at primary series and first booster, control vaccine at second and third booster, n = 400, 5-36 months olds.
  For the school age booster extension, group 3-1 has been randomised into two groups: group 5 and 6. Group 5 will receive another dose of R21/Matrix-M.
  Interventions: Biological: R21/Matrix-M; Biological: Rabies vaccine, Hepatitis A vaccine or Meningococcal vaccine
- Seasonal Regime - Group 3-2 (Experimental): R21/Matrix-M at primary series, first booster and second booster, control vaccine at third booster, n = 400, 5-36 months olds.
  For the school age booster extension, this group will receive no further vaccination and will be followed up for a further two years.
  Interventions: Biological: R21/Matrix-M; Biological: Rabies vaccine, Hepatitis A vaccine or Meningococcal vaccine
- Seasonal Regime - Group 3-3 (Experimental): R21/Matrix-M at primary series and first booster, control vaccine at second booster and R21/Matrix-M at third booster, n = 400, 5-36 months olds.
  For the school age booster extension, this group will receive no further vaccination and will be followed up for a further two years.
  Interventions: Biological: R21/Matrix-M; Biological: Rabies vaccine, Hepatitis A vaccine or Meningococcal vaccine
- Seasonal Regime - Group 3-4 (Experimental): R21/Matrix-M at primary series, first booster, second booster and third booster, n = 400, 5-36 months olds.
  For the school age booster extension, this group will receive no further vaccination and will be followed up for a further two years.
  Interventions: Biological: R21/Matrix-M
- Seasonal Regime - Group 4 (Placebo Comparator): Control vaccine at primary series, first booster, second booster and third booster, n=800, 5-36 month olds.
  For the school age booster extension, this group will receive one further booster of the control vaccine.
  Interventions: Biological: Rabies vaccine, Hepatitis A vaccine or Meningococcal vaccine
- Seasonal Regime - Group 6 (Experimental): Group 3-1 for the initial part of the trial and first extension - R21/Matrix-M at primary series and first booster, control vaccine at second and third booster, n = 400, 5-36 months olds.
  For the school age booster extension, group 3-1 has been randomised into two groups: group 5 and 6. Group 6 will receive a control vaccine.
  Interventions: Biological: R21/Matrix-M; Biological: Rabies vaccine, Hepatitis A vaccine or Meningococcal vaccine

INTERVENTIONS:
Biological: R21/Matrix-M — Adjuvanted malaria vaccine
  Arms: Seasonal Regime - Group 3-2; Seasonal Regime - Group 3-3; Seasonal Regime - Group 3-4; Seasonal Regime - Group 5; Seasonal Regime - Group 6; Standard Regime - Group 1-1; Standard Regime - Group 1-2; Standard Regime - Group 1-3; Standard Regime - Group 1-4
Biological: Rabies vaccine, Hepatitis A vaccine or Meningococcal vaccine — Placebo Comparator
  Arms: Seasonal Regime - Group 3-2; Seasonal Regime - Group 3-3; Seasonal Regime - Group 4; Seasonal Regime - Group 5; Seasonal Regime - Group 6; Standard Regime - Group 1-1; Standard Regime - Group 1-2; Standard Regime - Group 1-3; Standard Regime - Group 2

SUMMARY:
A Phase III randomized controlled multi-centre trial to evaluate the efficacy of the R21/Matrix-M vaccine in African children against clinical malaria

DETAILED DESCRIPTION:
This will be a double-blind, individually randomised trial. In the first phase of the trial, participants were randomised 2:1 to receive R21/Matrix-M malaria vaccine or a control rabies vaccine (Abhayrab). The study groups are as follows:

Standard vaccination regime, 5-36 months olds R21/Matrix-M x 3, n = 1600 Control (rabies) vaccine x 3, n = 800

Seasonal vaccination regime, 5-36 month olds R21/Matrix-M x 3, n = 1600 Control (rabies) vaccine x 3, n = 800

In each group, a booster (4th) dose of the same vaccine will be administered 12 months after the third dose. At certain trial sites, participants in the malaria vaccine group may be further randomised 1:1 to receive a single-vial: two-vial formulation of R21/Matrix-M.

The trial has been extended for two further years to assess safety and efficacy over a longer period of time. During this time, it will also assess the safety, immunogenicity and efficacy of second and third booster doses.

One year after the first booster (fourth dose), participants in the R21/Matrix-M arm will be further randomised 1:1:1:1 to four groups to receive:

1. No booster doses (total of 4 doses of R21/Matrix-M).
2. One booster dose, one year after the first booster dose (total of 5 doses of R21/Matrix-M)
3. One booster dose, two years after the first booster dose (total of 5 doses of R21/Matrix-M)
4. Two booster doses, one year apart (total of 6 doses of R21/Matrix-M)

Participants who are not receiving R21/Matrix-M, will receive a control vaccine at the relevant time point of vaccine administration The control vaccine for the second and the third booster will be a licensed Hepatitis A vaccine.

Participants will be followed up for 12 months after their third booster.

2400 participants will be enrolled for the standard vaccination regime in: Dande, Burkina Faso; Kilifi, Kenya; and Bagamoyo, Tanzania.

In addition, a further 2400 participants will be enrolled for the seasonal vaccination regime in Nanoro, Burkina Faso and Bougouni, Mali.

Study population

Standard vaccination regime:

5-36 month old children living permanently in the study area who are eligible.

Seasonal vaccination regime:

5-36 month old children living permanently in the study area who are eligible.

Primary study objectives

Efficacy:

* To assess the protective efficacy of R21/Matrix-M against clinical malaria caused by Plasmodium falciparum, in 5-36 month old children living in a malaria endemic area, 12 months after completion of the primary course (standard vaccination regime).
* To assess the protective efficacy of R21/Matrix-M against clinical malaria caused by Plasmodium falciparum, in 5-36 month old children living in a malaria endemic area, 12 months after completion of the primary course (seasonal vaccination regime).

Safety:

• To assess the safety and reactogenicity of R21/Matrix-M, in both vaccination regimes, of children living in a malaria endemic area, in the month following each vaccination, and 12 months after completion of the primary course.

Secondary objectives

* Efficacy against clinical malaria after each booster vaccination
* Efficacy against clinical malaria after the primary series and booster vaccination, regardless of vaccination regime
* Efficacy against asymptomatic P. falciparum infection.
* Efficacy against severe malaria disease.
* Efficacy according to different transmission settings.
* Efficacy against incident severe anaemia, blood transfusion requirement and malaria hospitalisation.
* Safety and reactogenicity (including Serious adverse events (SAEs) and any deaths) following each booster vaccination and for the duration of the study.
* Assessment of humoral immunogenicity by anti-CSP antibody concentrations measured 12 months after completion of the primary series of 3 vaccinations and 12 months after booster vaccinations.
* Safety, immunogenicity and efficacy of a single- vial formulation of R21/Matrix-M

This trial is funded by the Serum Institute of India.

The trial has been extended in 2025 for a further two years in both seasonal sites (Nanoro, Burkina Faso and Bougouni, Mali) when children will be of school age.

In this extension, participants who received 4 doses of R21/Matrix-M in the previous part of the trial will be randomised to receive a 5th dose of R21/Matrix-M or a control vaccine and will be followed up for 2 years. Participants in the control group from the previous part of the trial will receive one dose of a control vaccine and will be followed up for 2 years. Participants who have received 5 or 6 doses of R21/Matrix-M will not receive further vaccinations but will be followed up for two more years, (a total of 3 years since the last vaccination (R21/Matrix-M or control vaccine)).

ELIGIBILITY:
Inclusion Criteria:

All participants must satisfy the following criteria at study entry:

* The child is 5-36 months of age at the time of first vaccination.
* Signed informed consent/thumb-printed and witnessed informed consent obtained from the parent(s)/guardian(s) of the child to join the trial.
* The investigator believes that the parents/guardians can and will comply with the requirements of the protocol if the child is enrolled in the study.
* The child is a permanent resident of the study area and likely to remain a resident for the duration of the trial.

Exclusion Criteria:

The following criteria should be checked at the time of study entry. If any apply, the participant must not be included:

* The child has previously received a malaria vaccine.
* The child is enrolled in another malaria intervention trial.
* The child has a history of allergic disease or reactions likely to be exacerbated by any component of the malaria or control vaccine.
* The child has a history of allergic reactions, significant IgE-mediated events or anaphylaxis to previous immunisations.
* The child has major congenital defects.
* The child has anaemia associated with clinical signs of symptoms of decompensation, or a haemoglobin of ≤ 5.0 g/dL.
* The child has had a blood transfusion within one month of enrolment.
* The child has been administered immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate.
* The child has malnutrition requiring hospital admission.
* The child has an acute or chronic, clinically significant pulmonary, cardiovascular, gastrointestinal, endocrine, neurological, skin, hepatic or renal functional abnormality, as determined by medical history, physical examination or laboratory tests.
* Children currently meeting the WHO criteria for HIV disease of stage 3 or 4 severity. A previous history of stage 3 or 4 disease is not an exclusion. Note: There will be no routine testing for HIV. Positive diagnoses will be recorded at screening if known.
* The child has received an investigational drug or vaccine other than the study vaccines within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* The child is currently participating in another clinical trial if likely to affect data interpretation of this trial
* The child has any significant disease, disorder or situation which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.

Additional exclusion criteria for second phase of the trial (addition of second and third booster doses)

- Hypersensitivity to neomycin (Hepatitis A vaccine may contain traces of this).

Ages: 5 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 4800 (Estimated)
Dates: Start 2021-04-29 (Actual); Primary Completion 2023-03-21 (Actual); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Efficacy: To assess the protective efficacy of R21/Matrix-M against clinical malaria caused by Plasmodium falciparum, in 5-36 month old children living in a malaria endemic area, 12 months after completion of the primary course. | 2 years
  The primary efficacy outcome is clinical malaria, according to the primary case definition: the presence of axillary temperature ≥37.5°C and/ or history of fever within the last 24 hours, and P. falciparum asexual parasitaemia >5000 parasites/μL.This will assessed separately for seasonal and standard vaccination regimes.
Safety: To assess the safety and reactogenicity of R21/Matrix-M, in both vaccination regimes, of children living in a malaria endemic area, in the month following each vaccination, and 12 months after completion of the primary course. | 2 years
  * Occurrence of solicited local reactogenicity signs and symptoms for 7 days following the vaccination.
  * Occurrence of solicited systemic reactogenicity signs and symptoms for 7 days following the vaccination.
  * Occurrence of unsolicited adverse events for 28 days following the vaccination.
  * Change from baseline for safety laboratory measures thought to be clinically significant.
  * Occurrence of serious adverse events for the whole study duration.
School age booster extension: To assess the protective efficacy of R21/Matrix-M against clinical malaria caused by Plasmodium falciparum in school- age children in Burkina Faso and Mali | 12 months and 24 months after school age booster
  * To assess the protective efficacy of an additional late booster of R21/Matrix-M at 24 months against clinical malaria, in school-age children who have previously received four doses of R21/Matrix-M.
  * To assess the protective efficacy of R21/Matrix-M at 24 months against clinical malaria, in school- age children, who have previously received four doses of R21/Matrix-M.
  * To assess the protective efficacy of R21/Matrix-M at 12 months against clinical malaria, in school- age children, who have previously received a fifth dose one year after the fourth dose, a delayed fifth dose or six doses of R21/Matrix-M.
  * To assess the protective efficacy of R21/Matrix-M at 12 months against clinical malaria, in school- age children who have previously received a fifth dose one year after the fourth dose, a delayed fifth dose or six doses of R21/Matrix-M compared to those who received 4 doses.
School age booster extension: to assess the safety and reactogenicity of an additional late booster of R21/Matrix-M, in school age children living in Burkina Faso and Mali, one month after vaccination | One month after the school age booster
  This will be measured through the occurrence of local and systemic reactogenicity signs and symptoms for 7 days following the school age booster, and the occurrence of unsolicited adverse events for 28 days following this booster.

SECONDARY OUTCOMES:
Protective efficacy of R21/Matrix-M against clinical malaria caused by P.falciparum, in 5-36 month old children living in a malaria endemic area, following the primary vaccination series across both vaccination regimes and following booster vaccinations. | 2 years
  * Efficacy against clinical malaria following the primary series, regardless of vaccination regime.
  * Efficacy against clinical malaria after each booster vaccination. This will be assessed for the seasonal vaccination regime, standard vaccination regime and across both vaccination regimes together.
  Clinical malaria is defined (according to the primary case definition) as the presence of axillary temperature ≥37.5°C and/ or history of fever within the last 24 hours, and P. falciparum asexual parasitaemia >5000 parasites/μL.
Efficacy of R21/Matrix-M against asymptomatic P.falciparum malaria infection in either vaccination regime, following the primary vaccination series and following each booster vaccination. | 2 years
  Asymptomatic malaria, defined by: Presence of axillary temperature <37.5°C and absence history of fever within the last 24 hours AND P. falciparum asexual parasitaemia > 0 parasites/μL.
Efficacy of R21/Matrix-M against severe malaria disease in either vaccination regime, following the primary vaccination series and following each booster vaccination. | 2 years
  Severe malaria, defined by the primary case definition:
  Presence of P. falciparum asexual parasitaemia > 5000 parasites/μL
  AND one of more of the following criteria of disease severity:
  * Prostration
  * Respiratory distress
  * Blantyre coma score ≤ 2
  * Seizures: 2 or more
  * Hypoglycaemia < 2.2 mmol/L
  * Acidosis BE ≤-10.0 mmol/L
  * Lactate ≥ 5.0 mmol/L
  * Anaemia < 5.0 g/dL AND without any of the following diagnosis of co-morbidity
  * Pneumonia (confirmed by X-ray)
  * Meningitis (confirmed by Cerebrospinal Fluid examination)
  * Sepsis (with Positive blood culture)
  * Gastroenteritis with dehydration
Efficacy of R21/Matrix-M against clinical malaria according to different transmission settings (seasonal and standard vaccination regimes). | 2 years
  Clinical malaria is defined (according to the primary case definition) as the presence of axillary temperature ≥37.5°C and/ or history of fever within the last 24 hours, and P. falciparum asexual parasitaemia >5000 parasites/μL.
Efficacy of R21/Matrix-M against incident severe anaemia and the need for blood transfusion in both vaccination regimes following the primary vaccination series and each booster vaccination. | 2 years
  Incident severe anaemia according to the primary case definition: Documented Hb <5.0 g/dL identified at clinical presentation in association with P. falciparum asexual parasitaemia > 5000 parasites/μL.
  Incident severe anaemia according to the secondary case definitions:
  * Documented Hb <5.0 g/dL identified at clinical presentation in association with P. falciparum asexual parasitaemia > 0 parasites/μL
  * Documented Hb <5.0 g/dL identified at clinical presentation and requirement for a blood transfusion
  * Documented Hb <5.0 g/dL identified at clinical presentation
  Prevalent severe anaemia defined as: Documented Hb <5.0 g/dL
  Prevalent moderate anaemia defined as: Documented Hb <8.0 g/dL
  Prevalent mild anaemia defined as: Documented Hb <10.0 g/dl
Efficacy of R21/Matrix-M against malaria hospitalisation following the primary vaccination series and each booster vaccination. | 2 years
  Malaria hospitalisation defined by the primary case definition: Medical hospitalisation with confirmed P. falciparum asexual parasitaemia > 5000 parasites/μL.
  Malaria hospitalisation defined by the secondary case definition: Medical hospitalisation which, in the judgement of the principal investigator, P. falciparum was the sole reason or major contributing factor.
Safety, reactogenicity, humoral immunogenicity and efficacy of R21/Matrix-M as a single-vial formulation, compared with the two-vial formulation. | 2 years
  Safety and reactogenicity of the single-vial formulation will be assessed as per the primary safety outcome (#2).
  Efficacy of the single-vial formulation will be assessed as per the primary efficacy outcome (#1).
  Immunogenicity will be assessed as per the secondary immunogenicity outcome (#11).
Safety and reactogenicity (including Serious adverse events (SAEs) and any deaths) following each booster vaccination and for the duration of the study. | 2 years
  Safety as per the primary outcome measures for safety but to be assessed post boost vaccinations.
Humoral immunogenicity by anti-CSP antibody concentrations measured 12 months after completion of the primary series of 3 vaccinations and 12 months after each booster vaccination. | 2 years
  * Comparison of immunogenicity (antibody responses to CSP) in the R21/Matrix-M vaccination groups with those in the control vaccine groups and the durability of responses
  * Serology to quantify antibodies to the vaccine components (regions of the CS antigen including the NANP repeat region and other elements of the protein as well as antibodies to HBsAg).
School age booster extension: Efficacy | 6, 12, 18 and 24 months after receiving a school age booster
  * Efficacy against clinical malaria at 6, 12 and 18 months after receiving a school age booster.
  * Efficacy against asymptomatic P. falciparum infection at 6, 12, 18 and 24 months after receiving a school age booster.
  * Efficacy against severe malaria disease at 12 and 24 months after receiving a school age booster.
  * Efficacy against severe anaemia at 12 and 24 months after receiving a school age booster.
School age booster extension: Safety and reactogenicity | Two years after school age booster
  Safety and reactogenicity (including Serious adverse events (SAEs) and any deaths) following the school age booster vaccination and for the duration of the study.
School age booster: Immunogenicity | 28 days post school age booster, 1 year post school age booster and 2 years post school age booster
  * To evaluate immunogenicity, magnitude, quality and functionality of induced antibodies to the circumsporozoite protein, antibodies to HBsAg and other exploratory immunological endpoints in all vaccination groups.
  * To assess vaccine-induced potential immune correlates of vaccine efficacy.
School age booster extension: Impact | 2 years after school age booster
  * Assessment of impact of a school age booster of R21/Matrix-M on school attendance.
  * Assessment of public health impact and cost-effectiveness of a school-age booster through modelling.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian VS Hill, PhD, Principal Investigator — Jenner Institute, University of Oxford
Locations (1):
- CCVTM, University of Oxford, Churchill Hospital, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Datoo MS, Dicko A, Tinto H, Ouedraogo JB, Hamaluba M, Olotu A, Beaumont E, Ramos Lopez F, Natama HM, Weston S, Chemba M, Compaore YD, Issiaka D, Salou D, Some AM, Omenda S, Lawrie A, Bejon P, Rao H, Chandramohan D, Roberts R, Bharati S, Stockdale L, Gairola S, Greenwood BM, Ewer KJ, Bradley J, Kulkarni PS, Shaligram U, Hill AVS; R21/Matrix-M Phase 3 Trial Group. Safety and efficacy of malaria vaccine candidate R21/Matrix-M in African children: a multicentre, double-blind, randomised, phase 3 trial. Lancet. 2024 Feb 10;403(10426):533-544. doi: 10.1016/S0140-6736(23)02511-4. Epub 2024 Feb 1. PMID 38310910